CLINICAL TRIAL: NCT05660902
Title: THE EFFECT OF EXERCISES ON FUNCTIONAL INDEPENDENCE AND QUALITY OF LIFE IN INDIVIDUALS WITH A STROKE
Brief Title: EFFECT OF EXERCISES IN PATIENTS WITH STROKE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Özlem Ceyhan, Principal Investigator, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: SVHROM
Record Dates: First submitted 2022-12-06; First posted 2022-12-21 (Actual); Last update posted 2022-12-21 (Actual); Status verified 2022-12

CONDITIONS: Stroke; Exercise
Keywords: Functional Independence; Stroke; ROM Exercises; Quality of Life
MeSH Terms: conditions — Stroke; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Patients in this group continued their routine medical treatment program without any treatment.
- Intervention Group (Experimental): Patients in this group continued their routine medical treatment program without any treatment. Moreover, ROM exercises were performed by the researcher and health personnel trained by the researcher 3 times a day for 2 weeks, approximately 30 minutes.
  Interventions: Other: ROM Exercises

INTERVENTIONS:
Other: ROM Exercises — The patients were evaluated by the physician, they were put into practice when their condition was stable within the first 72 hours. In addition to their routine treatments, according to the ROM exercise protocol, which was created by taking expert opinions and reviewing the literature ROM exercises were performed by the researcher and health personnel trained by the researcher 3 times a day for 2 weeks, approximately 30 minutes. The movements were started with the upper extremity on the unaffected side and then moved to the affected upper extremity. After the exercise applied to the affected upper extremity was finished, the same exercise was applied to the intact lower extremity and the affected lower extremity. Only the resistance points were mobilized and the exercise applied in each joint was repeated at least three times without applying extra force.
  Other Names: Intervention Group
  Arms: Intervention Group

SUMMARY:
Aim: This study was conducted as a randomized controlled experimental study to determine the effect of ROM exercises applied to individuals who had a stroke on functional independence and quality of life.

Design: This study was conducted as a randomized controlled experimental study Methods: The study was conducted with 80 individuals, 40 of whom were in the intervention group and 40 in the control group, who received inpatient treatment in the neurology service of a regional city hospital, and met the inclusion criteria. Planned ROM exercises were applied to the individuals in the intervention group 3 times a day for 2 weeks, and no application was made to the control group other than routine treatment. Data were collected by the researcher using the Questionnaire Form, Patient Information Form, Functional Independence Scale and Stroke Specific Quality of Life Scale.

ELIGIBILITY:
Inclusion Criteria:

* Being over 18 years old,
* Coming to the hospital within 72 hours of having a stroke,
* A definitive diagnosis of Cerebrovascular Diseases according to the diagnostic criteria,
* Having a hemiplegic condition,
* Having a score of 13 or higher on the Glasgow Coma Scale,
* Not to be involved in any special exercise program other than the service routine,
* Having approval from the clinician about there is no harm in doing ROM exercises,
* Agreeing to participate in the study

Exclusion Criteria:

* People with quadriplegia/tetraplegia,
* Those with psychiatric illnesses,
* Those who have any extremity amputated,
* Those who have open wounds that prevent exercise and cause bleeding,
* Those with fractures in their body and those who had an orthopedic operation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Stroke Specific Quality of Life Scale (SS-QOL) | When the first patient was included in the group.
  The scale, which has a total of 49 items, consists of questions evaluating mobility, energy, upper extremity functioning, self-care, work/productivity, mood, social roles, family roles, vision, language, thinking, and personality traits. The items on the scale are scored according to a five-point Likert scale: 1. strongly agree, 2. partially agree, 3. undecided, 4. partially disagree, 5. strongly disagree.
Stroke Specific Quality of Life Scale (SS-QOL) | İt was applied face-to-face at the end of the 2nd week
  The scale, which has a total of 49 items, consists of questions evaluating mobility, energy,
Stroke Specific Quality of Life Scale (SS-QOL) | When called for control at the end of the 4th week
  The scale, which has a total of 49 items, consists of questions evaluating mobility, energy,

SECONDARY OUTCOMES:
Functional Independence Measure (FIM) | When the first patient was included in the group.
  The scale consists of 6 functional sections: self-care, sphincter, transfer, locomotion, communication, and social cognition. In FIM, a total of 18 activities are evaluated for functional independence using a 7-point scale for each. Level 1 represents total assistance, and level 7 represents complete independence. The highest score that can be obtained in total is 126, and the lowest score is 18. There is a direct correlation between a high score and functional independence level
Functional Independence Measure (FIM) | İt was applied face-to-face at the end of the 2nd week
  The scale consists of 6 functional sections: self-care, sphincter, transfer, locomotion,
Functional Independence Measure (FIM) | When called for control at the end of the 4th week
  The scale consists of 6 functional sections: self-care, sphincter, transfer, locomotion,

CONTACTS AND LOCATIONS:
Locations (1):
- ERciyes University, Kayseri, Turkey (Türkiye)

REFERENCES:
- [Background] Munce SEP, Perrier L, Shin S, Adhihetty C, Pitzul K, Nelson MLA, Bayley MT. Strategies to improve the quality of life of persons post-stroke: protocol of a systematic review. Syst Rev. 2017 Sep 7;6(1):184. doi: 10.1186/s13643-017-0579-3. PMID 28882175
- [Background] Thommasen HV, Zhang W. Impact of chronic disease on quality of life in the Bella Coola Valley. Rural Remote Health. 2006 Apr-Jun;6(2):528. Epub 2006 Jun 5. PMID 16749870
- [Background] Young JA, Tolentino M. Neuroplasticity and its applications for rehabilitation. Am J Ther. 2011 Jan;18(1):70-80. doi: 10.1097/MJT.0b013e3181e0f1a4. PMID 21192249
- [Background] Xu BH, Yu RQ, Yu W, Xie B, Huang YX. [Effects of early rehabilitation on activities of daily living and complications in acute stroke patients]. Beijing Da Xue Xue Bao Yi Xue Ban. 2004 Feb;36(1):75-8. Chinese. PMID 14970894
- [Background] Wee HL, Cheung YB, Li SC, Fong KY, Thumboo J. The impact of diabetes mellitus and other chronic medical conditions on health-related Quality of Life: is the whole greater than the sum of its parts? Health Qual Life Outcomes. 2005 Jan 12;3:2. doi: 10.1186/1477-7525-3-2. PMID 15644146